CLINICAL TRIAL: NCT00502450
Title: Is There Hearing Loss After Acute Mastoiditis
Status: Withdrawn | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: eyal raveh, schneider
Other Study IDs: 4560
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2007-07

CONDITIONS: Acute Mastoiditis; Acute Otitis Media
Keywords: Acute mastoiditis; Hearing loss; Mastoidectomy; Audiogram
MeSH Terms: conditions — Otitis Media; Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
Following acute mastoiditis there is a possible risk to develop hearing loss. The cause could be either possible involvement of the inner ear, or in cases that underwent surgery, secondary to the effect of the drill's noise. Extended hearing test will be performed for 25 children that suffered acute mastoiditis that resolved with conservative treatment and compared with 25 children that needed surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of acute mastoiditis 4 years and older

Exclusion Criteria:

* Younger than 4 years old Not cooperative for hearing test Active ear disease Major medical illness

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Raveh, MD, Study Director — Rabin Medical Center
Locations (1):
- Schneider Children'S Hospital, Petah Tikva, Israel